CLINICAL TRIAL: NCT01776359
Title: Effects of High Protein Intake With Intense Exercise and Energy Deficit
Acronym: RIPPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart M. Phillips, PhD, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: REB 12-670
Record Dates: First submitted 2013-01-14; First posted 2013-01-28 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Overweight
Keywords: Muscle; Protein; Diet; Exercise
MeSH Terms: conditions — Overweight; Motor Activity | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Protein (Active Comparator): High Protein
  Interventions: Dietary Supplement: High Protein
- Low Protein (Placebo Comparator): Low Protein
  Interventions: Dietary Supplement: Low Protein

INTERVENTIONS:
Dietary Supplement: High Protein — 2.4g/kg of protein
  Arms: High Protein
Dietary Supplement: Low Protein — 1.2g/kg of protein
  Arms: Low Protein

SUMMARY:
A four week intervention will take place with the participants. They will undergo 6 days a week of high intensity training. They will also be at a 40% energy deficiency. One group will have a normal intake of protein, 1.2g/kg, while the other will have 2.4g/kg. It is our thesis that the participants with the higher protein will retain more lean mass.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 males
* Healthy

Exclusion Criteria:

* more than 15% body fat
* 35-50ml/kg/min VO2
* BMI grater than 27

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Body Composition | 4 weeks
  To compare the effect of normal protein intake (1.2 g/kg per day) and increased protein intake (2.4 g/kg per day) on body composition over a 4 week period of energy restriction in young males (18-30), with intense exercise training. Body composition will be measured via DXA, Bod Pod, Bio-impedance, skin folds.

SECONDARY OUTCOMES:
Psychological state | 4 weeks
  To compare the psychological state of the participants, before, during and after the intervention. To see if the mind will grow with the body as high intensity exercise is performed, or whether the mind will tire and scores will be reduced. Measurement tactics will in include POMS, and PANAS questionnaires for mood, and stroop, isometric hand grip, operation span test, and vigilance task.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Mettler S, Mitchell N, Tipton KD. Increased protein intake reduces lean body mass loss during weight loss in athletes. Med Sci Sports Exerc. 2010 Feb;42(2):326-37. doi: 10.1249/MSS.0b013e3181b2ef8e. PMID 19927027
- [Background] Demling RH, DeSanti L. Effect of a hypocaloric diet, increased protein intake and resistance training on lean mass gains and fat mass loss in overweight police officers. Ann Nutr Metab. 2000;44(1):21-9. doi: 10.1159/000012817. PMID 10838463
- [Background] Butterfield GE, Calloway DH. Physical activity improves protein utilization in young men. Br J Nutr. 1984 Mar;51(2):171-84. doi: 10.1079/bjn19840021. PMID 6704368
- [Derived] Longland TM, Oikawa SY, Mitchell CJ, Devries MC, Phillips SM. Higher compared with lower dietary protein during an energy deficit combined with intense exercise promotes greater lean mass gain and fat mass loss: a randomized trial. Am J Clin Nutr. 2016 Mar;103(3):738-46. doi: 10.3945/ajcn.115.119339. Epub 2016 Jan 27. PMID 26817506